CLINICAL TRIAL: NCT00504738
Title: Evaluation of the Lungs of Individuals With Lung Disease With Segmental Bronchopulmonary Lung Lavage, Bronchial Brushing, and Bronchial Wall Biopsy (Qatar)
Brief Title: Lung Disease Collection (Qatar): Evaluation of the Lungs of Individuals With Lung Disease
Acronym: Q-LD
Status: Completed | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Weill Cornell Medical College in Qatar (Other); Hamad Medical Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 0604008489; HMC RC392/2006 (Other: Hamad Medical Corporation)
Record Dates: First submitted 2007-07-19; First posted 2007-07-20 (Estimated); Last update posted 2015-04-21 (Estimated); Status verified 2015-04

CONDITIONS: Lung Disease; Chronic Obstructive Pulmonary Disease (COPD); Asthma
Keywords: lung disease; chronic obstructive pulmonary disease (COPD); asthma; smokers; non-smokers
MeSH Terms: conditions — Lung Diseases; Pulmonary Disease, Chronic Obstructive; Asthma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The purpose of this protocol is to obtain biologic samples from the blood and lungs from patients with lung diseases in order to study the causes and indications of these disorders, learn how these lung disease manifest and progress, and how the lung disease can be treated.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this protocol is to obtain biologic samples from the blood and lungs from patients with lung diseases in order to study the causes and indications of these disorders, learn how these lung disease manifest and progress, and how the lung disease can be treated.

DETAILED DESCRIPTION:
The lung diseases are disorders associated with functional and/or structural derangements to the alveolar structures, airways, pulmonary blood vessels, pleura and/or mediastinum. The purpose of this protocol is to obtain biologic materials from the blood and lungs from these patients in order to: (1) develop an understanding of the etiology and pathogenesis of these disorders; and (2) identify individuals who will be suitable candidates for other protocols such as those involving investigational new drugs. As such, this protocol is part of the "infrastructure" for all of our human lung-related studies such as genomic/gene expression studies of airway epithelium and alveolar macrophages in all individuals with chronic obstructive lung disease (COPD), asthma, bronchogenic carcinoma, and pulmonary fibrosis compared to normal non-smokers and smokers, and studies of mediators in bronchoalveolar lavage fluid.

This protocol, to be carried out at Weill Cornell Medical College - Qatar and Hamad Medical Corporation, Qatar, parallels a similar approved protocol IRB #0005004440, entitled, "Evaluation of the Lungs of Individuals with Lung Disease with Segmental Bronchopulmonary Lung Lavage, Bronchial Brushing, and Bronchial Wall Biopsy", ongoing at Weill Cornell Medical College - New York.

ELIGIBILITY:
Inclusion Criteria:

Inclusion/Exclusion criteria for Part A

* Must provide informed consent
* Males and females, age 18 years and older
* Evidence of lung disease by at least one of the following:

  1. symptoms consistent with pulmonary disease;
  2. chest X-rays and/or chest CT consistent with lung disease;
  3. pulmonary function tests consistent with lung disease;
  4. lung biopsy consistent with lung disease;
  5. family history of lung disease;
  6. diseases of organs with known association with lung disease; and
  7. individuals suspected of having lung disease based on history and/or physical examination
* Undergoing fiberoptic bronchoscopy as dictated by their standard clinical care

Exclusion Criteria:

* Patient refuses consent.

Patients enrolled in Part A of the protocol will not undergo screening procedures/tests. These patients are undergoing a fiberoptic bronchoscopy as dictated by their standard clinical care and additional samples will be taken for research purposes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Recruitment will be from the patients of the Hamad Medical Corporation and others as relevant. The source of potential subjects will be the population of potential subjects with lung disease, as defined by the elegibility criteria, in Qatar. Accrual will be random with no bias as to gender or racial/ethnic group.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2006-04; Study Completion 2007-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald G. Crystal, MD, Principal Investigator — Weill Cornell Medical College, New York and Qatar
Locations (1):
- Hamad Medical Corporation, Doha, Qatar